CLINICAL TRIAL: NCT01039337
Title: Conservative Treatment for Hip Osteoarthritis: Effect of Manual Treatment and Hip School on Pain, Disability and Quality of Life - a Single-blinded Randomized Controlled Trial
Brief Title: Conservative Treatment for Hip Osteoarthritis
Acronym: COHART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Institute of Chiropractic and Clinical Biomechanics (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other); Foundation for Chiropractic Research and Post Graduate Education (Other); Region of Southern Denmark (Other); The Danish Rheumatism Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COHART; CVK S-20080027
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis, Hip
Keywords: osteoarthritis; manual therapy; manipulation; hip school; chiropractic; patient education
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hip school (Active Comparator): This group will receive hip school during the intervention period of 6 weeks.
  Interventions: Other: Hip School
- Hip School and Manual Treatment (Active Comparator): This group receives both hip school and manual treatment during the 6 weeks.
  Interventions: Other: Hip School and Manual Treatment
- Minimal control intervention (Active Comparator): An information leaflet including exercises.
  Interventions: Other: Minimal control intervention

INTERVENTIONS:
Other: Hip School — The hip school consists of one initial personal interview, three group sessions, and one follow-up personal interview. The hip school is a patient education programme which involves anatomy/physiology, epidemiology, disease progression and pain, advice on self-help and exercises.
  Arms: Hip school
Other: Hip School and Manual Treatment — Hip school as above. Patients receive manual treatment twice a week for 6 weeks. Manual treatment consists of joint manipulation and muscle energy techniques to the articular and soft-tissue structures of the hip.
  Arms: Hip School and Manual Treatment
Other: Minimal control intervention — As control group, an information leaflet is used with instructions to live as usual during the 6 weeks intervention period. The exercise sheet of the hip school is given to the patients with no further instruction.
  Arms: Minimal control intervention

SUMMARY:
The purpose of the study is to evaluate the effect of manual treatment and a patient education programme for patients without indication for hip surgery.

DETAILED DESCRIPTION:
Hip osteoarthritis (hip OA) is the second most common arthritis of the larger joints and may result in pain and disability and lead to reduced quality of life (QoL). The prevalence of hip OA, in the adult population, > 35 years, is estimated to 4-11% in the western society. In specific countries hip OA affects up to 25% in adults > 60 years. With a growing elder population, these prevalence rates will increase and the demand for cost-effective and safe interventions will increase as well.

International guidelines, 2008, on the management of hip and knee OA recommend a combination of non-pharmacological and pharmacological treatment. For years the majority of interventional research for hip and knee OA has focused on surgery and drugs. Surgery is an option, when pain and disability have reached severe levels, and an increasing group of patients are today looking for other treatment options than drug treatment (pharmacological). In the last 4-6 years, new randomized controlled trials (RCT) have shown promising results with non-pharmacological treatment, such as exercise, patient education, manual therapy and acupuncture.

The purpose of this RCT is to investigate the effect of combining manual treatment and a patient education programme and compare it to a minimal intervention in form of a home stretching programme. It will further investigate the specific effect of manual treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients referred from general practitioner, chiropractor or orthopaedic surgeon
* unilateral hip pain of minimum 3 months' duration
* radiology criteria for hip OA: joint space width (JSW) < 2.0 mm or a side difference in JSW of > 10%
* adequate mastering of the Danish language to complete instructions and questionnaires

Exclusion Criteria:

* inflammatory joint disease
* previous hip or knee alloplastic
* secondary arthritis due to hip fracture or infection
* bilateral hip pain
* hip dysplasia with a CE angle > 25 degrees and an AA angle > 10 degrees
* low back pain which dominates over the hip pain
* malignant disease
* patients with paresis or paralysis after neuromuscular, cerebrovascular or polyneuropathic disease
* hip pain resulting from labral tear, bursitis and/or snapping hip syndrome
* polyarthritis
* received manual treatment for the hip within the last year

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pain: Numerical pain scale | Baseline, 6 weeks, 3 months, 1 year

SECONDARY OUTCOMES:
Hip Disability and Osteoarthritis Outcome Score | Baseline, 6 weeks, 3 months, 1 year
General improvement experienced by patient - "Global Assessment" | Baseline, 6 weeks, 3 months, 1 year
Quality of life: EQ-5D | Baseline, 6 weeks, 3 months, 1 year
Passive hip range of motion | Baseline, 6 weeks, 3 months, 1 year
Hip surgery up to one year after baseline | Baseline, 6 weeks, 3 months, 1 year
Use of pain medication | Baseline, 6 weeks, 3 months, 1 year
Patient Specific Hip Disability | Baseline, 6 weeks, 3 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erik Poulsen, DC, MSc, Principal Investigator — Nordic Institute of Chiropractic and Clinical Biomechanics
Locations (1):
- Department of Ortopaedic Surgery and Traumatology, Odense University Hospital, Odense, DK, Denmark

REFERENCES:
- [Derived] Poulsen E, Hartvigsen J, Christensen HW, Roos EM, Vach W, Overgaard S. Patient education with or without manual therapy compared to a control group in patients with osteoarthritis of the hip. A proof-of-principle three-arm parallel group randomized clinical trial. Osteoarthritis Cartilage. 2013 Oct;21(10):1494-503. doi: 10.1016/j.joca.2013.06.009. Epub 2013 Jun 21. PMID 23792189
- [Derived] Poulsen E, Christensen HW, Roos EM, Vach W, Overgaard S, Hartvigsen J. Non-surgical treatment of hip osteoarthritis. Hip school, with or without the addition of manual therapy, in comparison to a minimal control intervention: protocol for a three-armed randomized clinical trial. BMC Musculoskelet Disord. 2011 May 4;12:88. doi: 10.1186/1471-2474-12-88. PMID 21542914